CLINICAL TRIAL: NCT06192134
Title: Continuous Passive Motion Device for Children With Arthrogryposis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Tariq Rahman, Principal Research Engineer, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1798457
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Arthrogryposis
MeSH Terms: conditions — Arthrogryposis

STUDY DESIGN:
Intervention Model Description: Pilot study of intervention compared to historic controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CPM group (Experimental): group receiving CPM therapy
  Interventions: Device: CPM device

INTERVENTIONS:
Device: CPM device — CPM brace

SUMMARY:
The Investigators are investigating a continuous passive motion device to exercise the knee of young children with arthrogryposis after they have had knee surgery.

DETAILED DESCRIPTION:
The investigators will measure the effect of continuous passive motion (CPM) of the knee joint post-surgery on young children with arthrogryposis. The investigators have developed a motorized brace that will move the joint through a prescribed range of motion and speed while the subject is seated. The objective of this pilot study is to develop the device from subject feedback and determine the right dose and speed of CPM to provide. CPM is routinely used for adults and older children after surgery to maintain range of motion. The machines used are too large for young children therefore the investigators have developed a prototype for small sized kids that will exercise their knee joint post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children with arthrogryposis
* Children between 3 and 7 years of age
* Children who have had recent knee surgery

Exclusion Criteria:

* Children older than 7
* Children unable to cooperate with protocol steps

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
range of motion | 2 weeks
  knee range of motion

IPD SHARING:
Plan to Share IPD: No